CLINICAL TRIAL: NCT06361953
Title: Comparing the Efficacy of Two Neurofeedback Protocols for Generalized Anxiety Disorder: Sensory Motor Rhythm and Alpha-Theta
Brief Title: Comparing the Efficacy of Two Neurofeedback Protocols for Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Abbas Masjedi Arani, Head of Clinical Psychology, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.SBMU.MSP.REC. 1401. 161
Record Dates: First submitted 2024-04-03; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alph-Theta (Experimental): 15 sessions of alpha (8-12Hz) and theta (4-8Hz) push on Pz based on 10-20 international system
  Interventions: Device: EEG Neurofeedback
- Sensory Motor Rhythm (Experimental): 15 sessions of sensory-motor rhythm (12-15Hz) push on Cz based on 10-20 international system
  Interventions: Device: EEG Neurofeedback

INTERVENTIONS:
Device: EEG Neurofeedback — neurofeedback training over five weeks, comprising 15 sessions. Each neurofeedback training session lasted 30 minutes.

SUMMARY:
Generalized anxiety disorder (GAD) is one of the most prevalent mental disorders in adults, marked by excessive and uncontrollable worry about various events or activities. It is accompanied by symptoms such as restlessness, irritability, fatigue, difficulty concentrating, problems with sleep, and somatic symptoms.

In addition, a critical and up-to-date comparison of different treatments for GAD is crucial due to their high costs and unsatisfactory outcomes. EEG neurofeedback training has not reached the same level of evidence as more extensively validated non-pharmacological treatments, such as cognitive behavioral therapy.This study aimed to compare the efficacy of two protocols: one targeting alpha-theta amplitude increase and the other concentrating on SMR.

ELIGIBILITY:
Inclusion Criteria:

* Normal hearing and vision,
* had never undergone neurofeedback sessions,
* diagnosed as GAD by a psychiatrist,
* no history of neurological disorders
* undergoing other therapies

Exclusion Criteria:

* started other treatments during the study
* missed more than one session

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
The Beck Anxiety Inventory | Pre-test, after 5 weeks and two month follow up
  higher scores mean higher depression
The Perceived Stress Questionnaire | Pre-test, after 5 weeks and two month follow up
  higher scores mean higher stress
Spielberger's state-trait anxiety test | Pre-test, after 5 weeks and two month follow up
  higher scores mean higher anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Beheshti University of Medical Science, Tehran, Iran